CLINICAL TRIAL: NCT01839071
Title: Influence of Vasculary Inflammation on Development of Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-077
Record Dates: First submitted 2013-03-21; First posted 2013-04-24 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease(CAD)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- biopsy of fat tissue (Other)
  Interventions: Procedure: biopsy

INTERVENTIONS:
Procedure: biopsy

SUMMARY:
The purpose of this study is to investigate if patients with coronary heart disease have higher risk to develop diabetes mellitus among the following two years.

The examination of biomarkers taken from blood and fat issue shall provide which factors could be responsible for development of diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* all patients with MI
* signed informed consent
* older than 18 years
* ability to give informed consent

Exclusion Criteria:

* absence of legal competence

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Fat tissue biopsy | 2 years
  Patients with Coronary artery disease(CAD) undergo a subcutane fat tissue biopsy to identify inflammation and diabetes biomarker, such as TNF, Adiponectin and Clock-Gene. This is done baseline, after 1 year and after 2 years. Comparison of the current measurements among the measurements of the following 2 years shall give evidence about the reasons and conditions of diabetes development.

SECONDARY OUTCOMES:
Blood collection | 2 years
  Blood of patients with Coronary artery disease(CAD)is taken to identify biomarkers of inflammation and diabetes, such as CRP, HbA1c, Adiponectin, Plasma MMp-9, s-ICAM-1, s-VCAM-1, P-selectin and Clock-Gene, CD11b/CD18, CD14, L-selectin, CD-64 and TNF. This is done baseline, after 1 year and after 2 years. Comparison of the current measurements among the measurements of the following 2 years shall give an evidence about the reasons and conditions of diabetes development.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Aachen, Aachen, North Rhine Westfalia, Germany